CLINICAL TRIAL: NCT04033081
Title: Registry of Retroperitoneal, Abdominal, Pelvic and Truncal Sarcoma Patients Treated With Permanently Implantable LDR CivaSheet® to Evaluate the Safety and Feasibility Over 5 Years
Brief Title: Registry of Sarcoma Patients Treated With Permanently Implantable LDR CivaSheet®
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CivaTech Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT007
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma
Keywords: CivaSheet; IORT; Intraoperative Radiation Therapy; Brachytherapy
MeSH Terms: conditions — Sarcoma | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CivaSheet Treatment (Experimental): Implanted with CivaSheet during tumor removal
  Interventions: Device: CivaSheet

INTERVENTIONS:
Device: CivaSheet — Implanting CivaSheet radiation therapy device at the time of surgery to irradiate surgical margin potentially preventing local recurrence
  Other Names: brachytherapy; Intraoperative Radiation Therapy

SUMMARY:
This patient study will determine the safety and toxicity of a permanently implantable brachytherapy source - CivaSheet® - which is designed to deliver a therapeutic dose of low dose rate (LDR) radiation with polymer encased Palladium-103. CivaSheet will be implanted in sarcoma patients with disease presenting in the retroperitoneum, abdomen, pelvis and trunk.

DETAILED DESCRIPTION:
CivaSheet® is an FDA-cleared product from CivaTech Oncology®. It is a series of small radioactive palladium-103 (Pd-103) sources on bio-absorbable, flexible, bio-compatible membrane. The CivaSheet can be custom cut in the operating room. The CivaSheet is 5 cm wide by 15 cm long and has a rim to allow an easy surface to suture. This flexible device can contour the surgical cavity delivering highly conformal and targeted radiation dose. CivaSheet can deliver a very high radiation dose to the surgical margin to potential prevent local cancer recurrence.

Sarcoma patients have up to 80% local recurrence rates, depending on histology and location of disease presentation. CivaSheet will be implanted at the surgical margin follow tumor removal. Monitoring the rate of acute toxicity is the primary endpoint. Secondary endpoints include disease progression and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

1. Subject Signed Inform Consent
2. Subject plans to remain in the long-term care of his/her enrolling center/investigators.
3. Sarcoma evident on imaging. Pathology biopsy proven or suspected by imaging but not a biopsy candidate.
4. Sarcoma in the retroperitoneum, abdomen, pelvis, or trunk
5. Subject is able to undergo surgery

Exclusion Criteria:

1. Is unable or unwilling to comply with protocol requirements.
2. Is enrolled in another study/registry not approved by CivaTech Oncology.
3. Pregnancy, breast feeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Rate of acute toxicity | 90 days post implant
  rate of greater than or equal to Grade 3 toxicity events based on CTCAE criteria

SECONDARY OUTCOMES:
Local control rate | 5 years
  rate of local tumor recurrences
Reoperation rate | 5 years
  Rate of re-operation for any reason
Complication rate | 6 months
  Rate of complications following device implant related or unrelated to the device
Dose to target and OAR | 90 days
  Amount of radiation dose delivered to the target volume and the adjacent organs at risk

CONTACTS AND LOCATIONS:
Overall Officials: Dian Wang, MD, Principal Investigator — Rush University Medical Center; Krisha Howell, MD, Principal Investigator — Michigan Healthcare Professionals
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No